CLINICAL TRIAL: NCT00211744
Title: Topiramate Augmentation in the Treatment of Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Ortho-McNeil Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Eric Hollander, Principal Investigator, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-0379
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Obsessive-compulsive Disorder
Keywords: OCD; Obsessive-Compulsive Disorder; OCD treatment
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
A 12-week program to examine the effectiveness of topiramate in adjunctive treatment for adults with obsessive-compulsive disorder and who are currently on serotonin reuptake inhibitor medications (ages 18-65).

DETAILED DESCRIPTION:
The Compulsive, Impulsive and Anxiety Disorders Program at the Mount Sinai School of Medicine is conducting a study of Topiramate (Topamax) added to an SSRI for the management of treatment-resistant Obsessive-Compulsive Disorder. The purpose of the study is to evaluate the safety and efficacy of Topiramate versus placebo added to a selective serotonin reuptake inhibitor (SRI) in patients with treatment resistant OCD. The program is 12 weeks in duration and involves regular visits with a psychiatrist as well as complete psychiatric and medical evaluations. Treatment and medication for the study will be provided free of charge.Participants must be between the ages of 18 and 65 and have an onset of OCD at least 1 year prior to screening. In addition, participants must be taking a clinically effective dose of an SSRI for at least 3 months and must maintain their current dose throughout the study. Participants must not have a primary OCD symptom of hoarding.

ELIGIBILITY:
Inclusion Criteria:

Males and Females 18-65 years of age diagnosed with OCD and currently taking SSRI medication(s)

Exclusion Criteria:

major medical disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2004-08; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of adjunctive topiramate vs. placebo in the treatment of OCD

CONTACTS AND LOCATIONS:
Overall Officials: Erik Hollander, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Berlin HA, Koran LM, Jenike MA, Shapira NA, Chaplin W, Pallanti S, Hollander E. Double-blind, placebo-controlled trial of topiramate augmentation in treatment-resistant obsessive-compulsive disorder. J Clin Psychiatry. 2011 May;72(5):716-21. doi: 10.4088/JCP.09m05266gre. Epub 2010 Aug 10. PMID 20816027